CLINICAL TRIAL: NCT06925620
Title: Effectiveness of Multimodal Information Technology-enhanced Hand Hygiene Improvement Strategy on Healthcare-associated Infections in Nursing Homes
Brief Title: Effectiveness of a Multimodal IT Enhanced Hand Hygiene Strategy on Healthcare Associated Infections in Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KMUHIRB-F(I)-20220007
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-03

CONDITIONS: Accuracy; Compliance; Healthcare-associated Infections
Keywords: Accuracy; Compliance; Density of Healthcare-Associated Infections; Information Technology; Knowledge; Multimodal Hand Hygiene Improvement Strategies; Nursing Homes
MeSH Terms: conditions — Patient Compliance; Cross Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): received a three-month IT-enhanced program.
  Interventions: Other: Multimodal Information Technology-based Hand Hygiene Strategies
- Control group (No Intervention): Continued routine care and only took part in the same measurements

INTERVENTIONS:
Other: Multimodal Information Technology-based Hand Hygiene Strategies — The intervention, adapted from the WHO's multimodal strategy, incorporated IT-based components to enhance hand hygiene compliance. A one-time, 1-hour online education session via Google Meet covered the WHO's Five Moments and seven-step handwashing technique, with real-time feedback using fluorescent dye and UV light. Post-session videos were available on tablets for review. Visual reminders, such as screensavers and digital posters, reinforced learning. Smart sanitizer dispensers with seven-step lights and a 20-second countdown were installed at five key sites, RFID-linked to staff badges for automatic tracking. Monthly performance data were shared via bulletin boards and LINE, with SMS feedback to top and bottom performers. Daily audio reminders played at 9 a.m. and 5 p.m., and high performers were recognized in monthly meetings.
  Arms: Experimental group

SUMMARY:
This study aims to evaluate the effectiveness of a multimodal hand hygiene improvement strategy, enhanced with information technology (IT), in reducing healthcare-associated infections (HAIs) in nursing homes. The goal is to improve infection prevention practices and promote a safer environment for older adults living in long-term care facilities.

DETAILED DESCRIPTION:
Hand hygiene is a key strategy for preventing healthcare-associated infections (HAIs), yet compliance among healthcare workers remains suboptimal due to knowledge gaps, limited resources, unfamiliarity with procedures, and poor adherence. This study aims to assess the effectiveness of an IT-enhanced multimodal hand hygiene intervention in reducing HAIs within nursing homes, thereby improving infection control practices and promoting a safer environment for older adults in long-term care settings.

ELIGIBILITY:
Inclusion Criteria:

* Full-time nurses or nursing assistants in the participating nursing homes
* Proficiency in Mandarin or Taiwanese

Exclusion Criteria:

• Confirmed or anticipated resignation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Hand Hygiene Knowledge | 1 month
  Cognitive scores were obtained through a "Hand Hygiene Knowledge Questionnaire for Long-term Care Facility Workers" It comprised 15 items (12 true/false, 2 multiple-choice, 1 multiple-answer), awarding 1 point for each correct answer and 0 for incorrect or unsure response, with a total score ranging from 0 to 15. Higher scores indicated greater hand hygiene knowledge.
Hand hygiene Compliance Rates | 4 month
  Hand hygiene compliance data were collected using the "Hand Hygiene Compliance Rate and Behavior Inspection Checklist for Long-term Care Facility Workers"(%)
Hand hygiene Accuracy Rates | 4 month
  Hand hygiene Accuracy data were collected using the "Hand Hygiene Compliance Rate and Behavior Inspection Checklist for Long-term Care Facility Workers"(%)
Density of healthcare-associated infections | 4 month
  A facility's "density of HAI" followed Taiwan's Centers for Disease Control (2012) guidelines(‰)

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Kaohsiung Nursing Home, Kaohsiung City
  - Pingtung Nursing Home, Pingtung City

IPD SHARING:
Plan to Share IPD: No
for personal privacy reason

DOCUMENTS (2):
  • Study Protocol (2022-01-27): https://cdn.clinicaltrials.gov/large-docs/20/NCT06925620/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-27): https://cdn.clinicaltrials.gov/large-docs/20/NCT06925620/SAP_001.pdf